CLINICAL TRIAL: NCT06099015
Title: Cera™ Vascular Plug System Post-Market Clinical Follow-Up: A Multi-center, Prospective, Observational, Single-arm, Open-label, Post-market Study
Brief Title: Cera™ Vascular Plug System Post-Market Clinical Follow-Up
Status: Recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LT-TS-22CE-04-01
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Aneurysm; Endoleak; Pulmonary Arteriovenous Malformation; Portal Hypertension; Arteriovenous Fistula; Splenic Laceration
Keywords: Lifetech; Cera Vascular Plug
MeSH Terms: conditions — Aneurysm; Endoleak; Pulmonary Arteriovenous Fistulas; Hypertension, Portal; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cera Vascular Plug Subjects: Patients who need arterial or venous embolization in the peripheral vasculature.
  Interventions: Device: Cera™ Vascular Plug System

INTERVENTIONS:
Device: Cera™ Vascular Plug System — The Cera™ Vascular Plug System is composed of Cera™ Vascular Plug and its accessory Introducer Kit. The Cera™ Vascular Plug is a self-expandable, cylindrical Ni-Ti wire mesh device.

SUMMARY:
The objective of the study is to collect and evaluate clinical data on patients of the Lifetech Cera™ Vascular Plug System to:

* confirm the performance
* confirm the safety
* identify previously unknown side-effects
* monitor the identified side-effects (related to the procedures or to the medical devices)
* identify and analyse emergent risks

DETAILED DESCRIPTION:
Lifetech Cera™ Vascular Plug System is indicated for arterial and venous embolization in the peripheral vasculature. This study, planned under the MDR requirements, aims to confirm the safety and performance of the Lifetech Cera™ Vascular Plug System, identify previously unknown side-effects, monitor the identified side-effects (related to the procedures or to the medical devices), identify and analyse emergent risks. The Study intends to enroll 132 subjects. The estimated enrollment period is 1 year, and the expected duration of each subject's participation is 1 year (i.e., the follow-up period). Final report shall be completed in 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 85;
2. Life expectancy > 1 year;
3. Require arterial or venous embolization in the peripheral vasculature;
4. Target embolization site(s) allow for safe insertion of the delivery catheter;
5. Voluntarily sign and date the Informed Consent Form (ICF) prior to any study-related activities commencement;
6. Willing and able to comply with protocol requirements, including all study visits and procedures.

Exclusion Criteria:

1. The subject is pregnant or plan to be pregnant or breast feeding;
2. The subject has a known allergy or hypersensitivity to any of the device materials including: nickel, stainless steel, polytetrafluoroethylene and titanium nitride;
3. The subject has a known allergy or hypersensitivity to contrast agent;
4. The subject has uncorrectable coagulopathy;
5. The subject has planned use of anticoagulant (e.g. direct thrombin inhibitors, factor Xa inhibitors, vitamin K antagonists) or antiplatelet therapy before, during and/or after treatment with the study device, which, in the opinion of the Investigator, would clinically interfere with the study endpoints
6. The subject has an unresolved systemic infection;
7. Subject who cannot tolerate general or local anesthesia;
8. The subject has a connective tissue disorders (e.g. Ehlers-Danlos Syndrome), arteritis (e.g. Takayasu's Disease) or another circulatory disorder;
9. The subject is participating in other drug or medical device clinical trials;
10. Any condition (medical or anatomic) making the subject not suitable for transcatheter embolotherapy according to the opinion of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need arterial or venous embolization in the peripheral vasculature.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Technical success | at procedure
  Complete occlusion of the target embolization site at the time of the procedure. A target embolization site is considered completely occluded if angiography showed no residual flow.

SECONDARY OUTCOMES:
Incidence of clinically relevant recanalization | at 3 months, 6 months, and 12 months post-procedure
  Clinically relevant recanalization is defined as recanalization through the study device that requires a re-intervention.
Incidence of clinically relevant migration | at 3 months, 6 months, and 12 months post-procedure
  Clinically relevant migration is defined as migration of the study device from the target embolization site that requires a re-intervention.
Incidence of device and/or procedure-related Adverse Events (AEs) | from attempted procedure to 12 months post-procedure
Incidence of device and/or procedure-related Serious Adverse Events (SAEs) | from attempted procedure to 12 months post-procedure
Incidence of device deficiencies | from attempted procedure to 12 months post-procedure
  Device deficiency means any inadequacy in the identity, quality, durability, reliability, safety or performance of an investigational device, including malfunction, use errors or inadequacy in the information supplied by the manufacturer.
Time to occlusion | at procedure
  Defined as the time from the device placement to complete occlusion of the target embolization sites.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No